CLINICAL TRIAL: NCT07275086
Title: Therapeutic Outcomes of Using Complementary Hand-based Treatment in Diabetes (TOUCH-D): A Pilot Single-group Feasibility Study Evaluating Biological and Psychological Effects of Swedish Massage in Adults With Type 1 Diabetes.
Brief Title: Therapeutic Outcomes of Using Complementary Hand-based Treatment in Diabetes
Acronym: TOHCD-D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Peter Johansson, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-05625
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: All participants receive Swedish massage once weekly for five weeks. Pre-post within-group design to explore biological and psychological effects and study feasibility.
Masking Description: Open-label single-group pilot study; neither participants nor investigators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swedish Massage (Experimental): Participants receive Swedish massage once weekly for five consecutive weeks. Each session lasts 45-60 minutes and is delivered by a licensed massage therapist. Techniques include kneading, gliding, and tapping of soft tissues, focusing on the back, shoulders, and neck. The massage is designed to promote relaxation and modulate stress-related biological systems
  Interventions: Behavioral: Swedish massage

INTERVENTIONS:
Behavioral: Swedish massage — Participants receive Swedish massage once weekly for five consecutive weeks. Each 45-60-minute session is delivered by a licensed massage therapist using traditional Swedish techniques (kneading, gliding, and tapping) focusing on the back, shoulders, and neck. The intervention aims to promote relaxation and modulate stress-related biological systems. The study uses a single-group pre-post design to explore biological and psychological effects and feasibility.

SUMMARY:
This pilot study evaluates potential biological and psychological effects of Swedish massage in adults with type 1 diabetes. Massage may influence stress-related mechanisms, such as hypothalamic-pituitary-adrenal (HPA) axis activity and inflammation, which are linked to impaired insulin sensitivity and glycemic control. Twenty participants with type 1 diabetes will receive weekly 45-60-minute Swedish massage sessions for five weeks. Biological outcomes include HbA1c, fasting glucose, copeptin, hs-CRP, IL-6, and TNF-α. Glycemic variability will be assessed using continuous glucose monitoring (CGM). Psychological outcomes include perceived stress (PSS-10) and anxiety (GAD-7). The study aims to explore feasibility, acceptability, and preliminary within-group effects on stress regulation and glycemic balance

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with type 1 diabetes ≥ 1 year
* Able to attend two assessment visits at Vrinnevi Hospital
* Uses CGM or equivalent system
* Able to communicate in Swedish and provide consent

Exclusion Criteria:

* Severe diabetes complications (e.g., advanced neuropathy)
* Acute psychiatric disorder requiring treatment
* Contraindications to massage (e.g., thrombosis, fever, infection, recent surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of HbA1c (mmol/mol) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  This measure is part of the study's limited efficacy evaluation and is used to explore preliminary within-group changes in preparation for a future randomized trial.
  HbA1c (mmol/mol), measured from fasting blood samples. Lower values indicate improved glycemic control.
Concentration of Copeptin (pmol/L) | Baseline and within 7 days after final massage (5 weeks).
  Limited efficacy outcome assessing preliminary within-group changes related to physiological stress.
  Copeptin measured from fasting serum samples. Lower concentrations indicate reduced stress system activation.
Concentration of high-sensitivity C-reactive protein, hs-CRP (mg/L) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group inflammatory changes.
  Lower concentrations indicate reduced systemic inflammation
Concentration of Interleukin-6 (IL-6) (pg/mL) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group inflammatory changes.
  Lower IL-6 levels indicate reduced inflammatory activation.
Mean interstitial glucose (mmol/L) measured by continuous glucose monitoring (CGM) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group changes in glycemic control.
  Mean interstitial glucose derived from CGM. Lower values indicate improved glycemic control.
Glycemic variability (Coefficient of Variation, %), measured by CGM | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group changes in glycemic stability.
  Lower %CV indicates more stable glucose levels.
Time in Range (percentage of CGM readings between 3.9-10 mmol/L) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group glycemic control. Higher percentages indicate improved glucose regulation.
Score on the Perceived Stress Scale-10 (PSS-10) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group psychological changes.
  The PSS-10 is a 10-item scale ranging 0-40, with higher scores indicating greater perceived stress.
Score on the Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group psychological changes.
  The GAD-7 ranges 0-21, with higher scores indicating more severe anxiety.
Concentration of fasting plasma glucose (mmol/L) | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Limited efficacy outcome assessing preliminary within-group metabolic changes prior to a future randomized trial.
  Fasting plasma glucose (mmol/L), with lower values indicating improved glycemic control.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline and within 7 days after the final massage session (5 weeks).
  This measure is part of the study's limited efficacy evaluation and is used to explore preliminary within-group changes in preparation for a future randomized trial.
  Clinic systolic blood pressure (mmHg), measured in a seated position after rest according to standard procedures. Lower values indicate improved cardiovascular risk profile.
Change in Diastolic Blood Pressure | Baseline and within 7 days after the final massage session (5 weeks).
  This measure is part of the study's limited efficacy evaluation and is used to explore preliminary within-group changes in preparation for a future randomized trial.
  Clinic systolic diastolic pressure (mmHg), measured in a seated position after rest according to standard procedures. Lower values indicate improved cardiovascular risk profile.

OTHER OUTCOMES:
Exploratory Metabolic and Inflammatory Markers | Change from baseline to within 7 days after the fifth massage session (5 weeks).
  Additional biomarkers related to stress physiology, inflammation, or short-term glycemic control may be analyzed if relevant and assay-ready samples are available (e.g., additional cytokines, oxidative stress markers, or alternative glycemic indices). These outcomes are exploratory and not required for completion of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Johansson, Norrköping, Linköpings Universitet, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to the small sample size and sensitive clinical information. De-identified summary data may be available upon reasonable request to the principal investigator for research purposes.